CLINICAL TRIAL: NCT06160752
Title: A Multicenter, Open-label, First-in-Human Study of TYRA-200 in Advanced Intrahepatic Cholangiocarcinoma and Other Solid Tumors With Activating FGFR2 Gene Alterations (SURF-201)
Brief Title: Safety and Anti-Tumor Activity of TYRA-200 in Advanced Cholangiocarcinoma With Activating FGFR2 Gene Alterations
Acronym: SURF201
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tyra Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYR200-101
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced Cholangiocarcinoma; Intrahepatic Cholangiocarcinoma; Solid Tumor; Metastatic Cholangiocarcinoma
Keywords: FGFR2 gene activation; FGFR2 gene alterations; FGFR2 gene fusion/rearrangement; FGFR2 gene mutation; FGFR2 gene translocation; FGFR2; Fibroblast growth factor receptor 2 (FGFR2); Fibroblast growth factor receptor 2 alterations; locally advanced cancer; metastatic cancer; solid tumors; cholangiocarcinoma; intrahepatic cholangiocarcinoma; unresectable cholangiocarcinoma; metastatic cholangiocarcinoma; fibroblast growth factor receptor inhibitor
MeSH Terms: conditions — Cholangiocarcinoma; Acrocephalosyndactylia; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Part A and Part B (Experimental): TYRA-200 taken once daily by mouth in 28-day cycles
  Interventions: Drug: Phase 1 Part A - dose escalation TYRA-200 taken once daily by mouth in 28-day cycles; Drug: Phase 1 Part B - dose expansion TYRA-200 taken once daily by mouth in 28-day cycles

INTERVENTIONS:
Drug: Phase 1 Part A - dose escalation TYRA-200 taken once daily by mouth in 28-day cycles — TYRA-200 is an oral, novel potent FGFR 1/2/3 tyrosine kinase inhibitor that targets tumors that contain activating gene alterations of FGFR2.
Drug: Phase 1 Part B - dose expansion TYRA-200 taken once daily by mouth in 28-day cycles — TYRA-200 is an oral, novel potent FGFR 1/2/3 tyrosine kinase inhibitor that targets tumors that contain activating gene alterations of FGFR2.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), and preliminary antitumor activity of TYRA-200 in cancers with FGFR2 activating gene alterations, including unresectable locally advanced/metastatic intrahepatic cholangiocarcinoma and other advanced solid tumors.

DETAILED DESCRIPTION:
This is a single arm, multi-part, phase 1 clinical trial studying TYRA-200, a novel, potent fibroblast growth factor receptor (FGFR) 1/2/3 tyrosine kinase inhibitor, in unresectable locally advanced/metastatic intrahepatic cholangiocarcinoma and other advanced solid tumors with activating alterations in FGFR2. Part A is a dose escalation study in participants with any advanced solid tumor with FGFR/FGF pathway alterations who have exhausted approved standard therapies. Part A will evaluate the safety, tolerability, and PK of TYRA-200 to determine the optimal and maximum tolerated dose (MTD). Part B will evaluate the preliminary antitumor activity of TYRA-200 in participants with unresectable locally advanced/metastatic intrahepatic cholangiocarcinoma who have previously received an FGFR inhibitor and have FGFR2 kinase-domain mutations resistant to other FGFR inhibitors.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 Part A

* Men and women 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* Any histologically confirmed advanced solid tumor with FGFR/FGF pathway alterations including FGFR gene mutations, fusions, and amplifications, as well as gene amplifications of FGFR ligands, who have exhausted or refused approved standard therapies.
* Evaluable disease according to RECIST v1.1.

Phase 1 Part B

* Men and women 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤1.
* Histologically confirmed locally advanced/metastatic intrahepatic cholangiocarcinoma with a previously identified FGFR2 gene mutation or rearrangement.
* Must have received a prior FGFR inhibitor. Participants may have received more than 1 prior FGFR inhibitor.
* Presence of an FGFR2 kinase domain mutation that confers resistance to previous/other FGFR inhibitors; resistance mutations should be identified by a US Food and Drug Administration authorized/approved companion diagnostic or a Clinical Laboratory Improvement Amendments (CLIA) validated local test performed in a certified laboratory.
* At least 1 measurable lesion by RECIST v1.1.

Exclusion Criteria:

* Discontinued a prior anti-FGFR therapy due to significant toxicity, defined as hepatotoxicity ≥Grade 3 or any Grade 4 toxicity according to CTCAE v5.0.
* Has a serum phosphorus level > upper limit of normal (ULN) during screening that remains >ULN despite medical management.
* Any ocular condition likely to increase the risk of eye toxicity.
* History of or current uncontrolled cardiovascular disease.
* Active, symptomatic, or untreated brain metastases.
* Gastrointestinal disorders that will affect oral administration or absorption of TYRA-200.
* Females who are pregnant, breastfeeding, or planning to become pregnant and males who plan to father a child while enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Part A: To determine the maximum tolerated dose (MTD) of TYRA-200. | Initiation of study treatment through 28 Days
Phase 1 Part B: To determine the optimal dose of TYRA-200. | Initiation of study treatment through 28 days (up to approximately 18 months

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs) as a measure of safety and tolerability. | From day 1 treatment through 28-days post treatment (up to 2 years)
Frequency in changes in laboratory parameters and physical signs of toxicity. | From day 1 treatment through 28-days post treatment (up to 2 years)
Pharmacokinetics: maximum plasma concentration (Cmax). | From Day 1 through Cycle 3 Day 1 (each cycle is 28 days)
Pharmacokinetics: time to reach maximum plasma concentration (Tmax). | From Day 1 through Cycle 3 Day 1 (each cycle is 28 days)
Pharmacokinetics: area under the plasma concentration-time curve (AUC). | From Day 1 through Cycle 3 Day 1 (each cycle is 28 days)
Pharmacokinetics: half-life of Tyra-200 (t1/2). | From Day 1 through Cycle 3 Day 1 (each cycle is 28 days)
Overall response rate (ORR) defined as the proportion of participants with complete response (CR) or partial response (PR) as determined by the investigator using RECIST V1.1. | From enrollment, every 8 or 12 weeks (up to 2 years)
Duration of response defined as the time from the initial CR or PR to the time of relapse or death, whichever occurs first among participant with an objective response. | From enrollment, every 8 or 12 weeks (up to 5 years)
Disease control rate defined as the proportion of participants having a CR, PR or stable disease (SD) for >12 weeks. | From enrollment up to 5 years
Time to response defined as time to first CR or PR that is subsequently confirmed according to RECIST v1.1. | Up to 5 years
Progression-free survival defined as the time from the date of first study drug administration to the earliest date of documented disease progression or death. | From the date of the first dose of study drug until disease progression or death as assessed up to the last efficacy assessment for disease progression (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Warner, Study Chair — Tyra Biosciences, Inc
Locations (4):
- United States (4):
  - University of California San Francisco (UCSF), San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Ohio State University, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas